CLINICAL TRIAL: NCT01918293
Title: Self-Management Using Smartphone Application for Chronic Disease Care in Real siTuation (SMART-Asthma) in Adult
Brief Title: Self-Management Using Smartphone Application for Chronic Disease Care in Real siTuation (SMART-Asthma): Adult
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Jongha Park, Study principal investigator, Inje University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SMART-ASTHMA (ADULT)
Record Dates: First submitted 2013-08-06; First posted 2013-08-07 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: BRONCHIAL ASTHMA
Keywords: ASTHMA; SMARTPHONE APPLICATION
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMART arm (Experimental): Using smartphone application for control of asthma
  Interventions: Device: SMART ARM
- conventional arm (No Intervention): non-using smartphone application for control asthma

INTERVENTIONS:
Device: SMART ARM — The smartphone application for self-management of Asthma offers symptom diary, general information for asthma, the information of asthma drugs,the guideline for inhaler and the specific action plan according to daily symptom and FEV1.
  Other Names: SMART-Asthma
  Arms: SMART arm

SUMMARY:
Bronchial asthma is an chronic airway disease with bronchial hypersensitivity due to inflammation and bronchial muscle contraction. It can cause recurrent dyspnea, cough, wheezing and severe life-threatening attack and lower quality of life. In addition, it make large amount of socioeconomic loss as about 3.7 billion US dollars.

ELIGIBILITY:
Inclusion Criteria:

* using smartphone
* alleged bronchial asthma over 3months & positive of bronchodilator response test or bronchial provocation test

Exclusion Criteria:

* COPD
* active pulmonary TUBERCULOSIS
* Acute exacerbation within 4weeks
* severe psychological disorder
* severe systemic disease; severe LC, ESRD ...
* MALIGNANCY

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-09; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The efficacy of smartphone application for asthma control test (ACT)and quality of life | at least 2 times a week
  Using ACT and ALQL score (QoL), we will investigate the efficacy of smanrtphone application for control of asthma compared to smartphone app. using group and smartphone app. non-using group

SECONDARY OUTCOMES:
FEV1 (Forced expiratory volume in 1 second ) and FVC (Forced vital capacity) | at least 1 time a month
  Using spirometer to check the variation of FEV1,we will investigate the efficacy of smanrtphone application for control of asthma compared to smartphone app. using group and smartphone app. non-using group
Acute exacerbation of bronchial asthma | at least 1 time a week
  Using medical record and questionaire of acute exacerbation,we will investigate the efficacy of smanrtphone application for control of asthma compared to smartphone app. using group and smartphone app. non-using group

CONTACTS AND LOCATIONS:
Locations (1):
- Haeundae Paik Hospital, Busan, South Korea